CLINICAL TRIAL: NCT00187109
Title: A Phase I/II Trial of Recombinant Human Thrombopoietin in Children With Malignant Solid Tumors and Lymphoma Receiving Ifosfamide, Carboplatin and Etoposide
Brief Title: Recombinant Human Thrombopoietin in Children Receiving Ifosfamide, Carboplatin, and Etoposide Chemotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPO
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2007-05

CONDITIONS: Germ Cell Tumors; Hepatic Cancer; Neuroblastoma; Osteosarcoma; Rhabdomyosarcoma
Keywords: Thrombocytopenia; Platelets; Thrombopoietin
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal; Liver Neoplasms; Neuroblastoma; Osteosarcoma; Rhabdomyosarcoma; Thrombocytopenia; Jacobs syndrome | interventions — Thrombopoietin

INTERVENTIONS:
Drug: Recombinant Human Thrombopoietin

SUMMARY:
Life-threatening thrombocytopenia (low platelet count) and neutropenia (low white blood count) remain the major dose-limiting toxicities following chemotherapy treatment for cancer. The only remedy for thrombocytopenia at present is platelet transfusion, which is effective in preventing life-threatening hemorrhage, but may lead to other complications. Preclinical studies and studies in adults have shown recombinant human thrombopoietin (rhTPO) to be effective in stimulating platelet production. The initial phase of this trial will evaluate the safety of rhTPO use immediately after chemotherapy with ifosfamide, carboplatin, and etoposide in children with solid tumors and lymphomas. The second phase of the study will evaluate the effectiveness of rhTPO in decreasing the duration of low platelet count after chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent, refractory, or previously untreated malignant solid tumor or recurrent/refractory lymphoma for which Ifosfamide, Carboplatin, and Etoposide chemotherapy is the most appropriate treatment.
* Adequate liver and kidney function.
* Adequate performance status.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40
Dates: Start 2000-06; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of recombinant human thrombopoietin following chemotherapy which includes ifosfamide, carboplatin and etoposide for solid tumors and lymphoma.
To evaluate whether recombinant human thrombopoietin will reduce the time necessary for platelet counts to recover following chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Najat C. Daw, M.D., Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org